CLINICAL TRIAL: NCT04577040
Title: Safety and Efficacy of Tadalafil vs. Tadalafil With Sildosin in the Management of Moderately and Severely Symptomatic Patients of Prostatic Hyperplasia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Yaseen, Menoufia governorate, Menoufia University
Other Study IDs: 10-2020urol
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Safety and Efficacy of Tadalafil vs. Tadalafil With Sildosin in the Management of Moderately and Severely Symptomatic Patients of Prostatic Hyperplasia
MeSH Terms: interventions — Tadalafil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Tadalafil in moderate puts
  Interventions: Drug: Tadalafil 5mg
- 2: Tadalafil in severe puts
  Interventions: Drug: Tadalafil 5mg
- 3: Tadalafil with sildosin in moderate luts
  Interventions: Drug: Tadalafil 5mg
- 4: Tadalafil with sildosin in severe luts
  Interventions: Drug: Tadalafil 5mg

INTERVENTIONS:
Drug: Tadalafil 5mg — Drugs
  Other Names: Sildosin

SUMMARY:
To study Safety and efficacy of Tadalafil vs. Tadalafil with Sildosin in the management of moderately and severely symptomatic patients of prostatic hyperplasia

DETAILED DESCRIPTION:
Introduction Benign prostatic hyperplasia (BPH) is a common cause of lower urinary tract symptoms (LUTS) in middle-aged and elderly men, and the incidence rate of LUTS associated with BPH (LUTS/BPH) increases with age.

LUTS can be broadly grouped into: (i) storage symptoms, such as frequency, urgency, and nocturia (ii) voiding symptoms, such as intermittency, weak stream and straining, and (iii) post-micturition symptoms, such as a feeling of incomplete emptying and post micturition dribble.

For optimal management of LUTS/BPH, medications should be chosen based on age, disease progression, need for long-term management, and other clinical parameters.

Alpha 1 adreno-receptors antagonists (alpha 1 blockers) are proposed as first-line drug therapy for LUTS/BPH as these agents reduce the adrenergic tone of the smooth muscle within the prostate and bladder neck, thereby relieving the bladder outlet obstruction.

Tadalafil (phosphodiesterase type 5 [PDE-5] inhibitor) was approved for treating LUTS/BPH. The inhibition of PDE-5leads to accumulation of cyclic guanosine monophosphate in the smooth muscles of the prostate and urethra which causes their relaxation resulting in alleviation of the symptoms of LUTS/BPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be included in the study will be either:

  1. diagnosis of BPH based on abdominal ultrasound or digital rectal examination.
  2. Moderate IPSS Score between 8 : 19.
  3. severe IPSS Score between 20 : 35.
  4. post void volume > 100 c.
  5. prostate size 50 to 80 gm.
  6. 2 or more weeks of freedom or washout from any medications known to influence LUTS before enrollment.
  7. mental and physical capacity to understand and fill out the study questionnaires.

Exclusion Criteria:

1. contraindications to Sildosin or Tadalafil.
2. diagnosis of prostate cancer.
3. possible presence of urinary infection, neurogenic bladder, stone bladder, refractory retention, hematuria of prostate origin or any cause for surgical intervention.
4. clinically significant cardiovascular, hepatic, or renal disorders.
5. cataract surgery planned during the study period.

Ages: 45 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Being in prostate patients
Study Population: Middle and old aged males
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Symptom relief | 2 weeks
  Decreased AUA score